CLINICAL TRIAL: NCT00874718
Title: Impact in Life Quality of a Educational Program for Prevention of Occupational Musculoskeletal Disorders in Workers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Antonio Cardoso dos Santos, Universidade Federal do Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2007755
Record Dates: First submitted 2009-03-31; First posted 2009-04-02 (Estimated); Last update posted 2009-04-02 (Estimated); Status verified 2009-03

CONDITIONS: Occupational Musculoskeletal Disorders; Healthy
Keywords: repetitive strain injury; quality of life; functional capacity; workers
MeSH Terms: conditions — Cumulative Trauma Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Action group (Active Comparator)
  Interventions: Behavioral: educational program
- Control group (Other): Non-specific educational program for general health.
  Interventions: Behavioral: General education

INTERVENTIONS:
Behavioral: educational program — 6-week educational program for prevention of occupational musculoskeletal diseases.
  Arms: Action group
Behavioral: General education — Non-specific educational program for general health.
  Arms: Control group

SUMMARY:
The study consists of evaluating the efficacy of an Educational Program for prevention of occupational musculoskeletal problems in workers. It is a randomized clinical trial with parallel groups and blinded evaluator, with a control group not submitted to the educational program, but that received a program for general orientation in health. The primary outcome was the change of the quality of life measured by means of Medical Outcomes Study 36-Term Short Health Survey (SF-36), that it is a generic instrument of evaluation of the quality of life, translated and validated in Portuguese of Brazil.

ELIGIBILITY:
Inclusion Criteria:

* All workers from a specific company, including administrative and production sections.

Exclusion Criteria:

* Workers absent from the workplace during all the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2007-10; Primary Completion 2008-08 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Medical Outcomes Study 36-Item Short Form Health Survey - (SF-36) | 6 months

SECONDARY OUTCOMES:
Work Limitation Questionnaire | 6 months
Work absenteeism | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo M Xavier, MD, Study Director — Associate Professor; Antonio C dos Santos, MD, Principal Investigator — Associate Professor
Locations (1):
- Federal University of Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Santos AC, Bredemeier M, Rosa KF, Amantea VA, Xavier RM. Impact on the Quality of Life of an Educational Program for the Prevention of Work-Related Musculoskeletal Disorders: a randomized controlled trial. BMC Public Health. 2011 Jan 28;11:60. doi: 10.1186/1471-2458-11-60. PMID 21276217